CLINICAL TRIAL: NCT02031718
Title: Comparison Between Interactive Internet-based Education and Counseling for the Management of Acne With That of Internet-based Education Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 511572
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online Education (No Intervention)
- Online Education & Virtual Counseling (Experimental): Online virtual counseling
  Interventions: Behavioral: Virtual Counseling

INTERVENTIONS:
Behavioral: Virtual Counseling
  Arms: Online Education & Virtual Counseling

SUMMARY:
This study will develop and evaluate the efficacy of an Internet-based education program incorporating virtual coaching. For this study, the virtual coach will consist of online videos aimed at providing acne education and promoting behaviors that support healthy skin. The use of Web-based technologies and virtual coaching in acne-related patient education is novel, and may significantly improve clinical outcomes and quality of life in acne patients. We hypothesize that an interactive Internet-based education and counseling program will be more effective than Internet-based education alone in improving clinical outcomes and quality of life in acne patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate acne vulgaris
* 13 years of age or older at time of assent, may be men or women.
* Able read and understand English.
* Able to hear and see the educational videos.
* Access to computer with Internet access.
* Capable of giving informed consent.
* Not currently using any prescription acne treatment.

Exclusion Criteria:

* Non-English speaking individuals.
* Self-reported exposure to environmental or chemical comedogenic agents
* Women with self-reported hyperandrogenism (e.g., PCOS)
* Women self-reporting current use of any form of specific acne-directed hormonal therapy
* Men or women with self-reported history of Cushing syndrome or congenital adrenal hyperplasia

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Acne Lesion Counts (Inflammatory and Non-inflammatory) | Up to 12 weeks

SECONDARY OUTCOMES:
Dermatology Life Quality Index | Up to 12 weeks

OTHER OUTCOMES:
Knowledge | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Wang, MD, Principal Investigator — University of California, Davis; April W Armstrong, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of California, Davis, Sacramento, California, United States

REFERENCES:
- [Derived] Tuong W, Wang AS, Armstrong AW. Effect of Automated Online Counseling on Clinical Outcomes and Quality of Life Among Adolescents With Acne Vulgaris: A Randomized Clinical Trial. JAMA Dermatol. 2015 Sep;151(9):970-5. doi: 10.1001/jamadermatol.2015.0859. PMID 26017816